CLINICAL TRIAL: NCT01441895
Title: A Post Market Pilot Study To Evaluate Corneal Sensation And The Incidence Of Dry Eye In Subjects Undergoing Refractive Cataract Extraction With The Femtosecond Laser For Arcuate Relaxing Incisions
Brief Title: Corneal Sensation and Incidence of Dry Eye Post Refractive Cataract Extraction With FemtoSecond Laser
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: AGN02-FEMTO
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Cataract; Dry Eye
Keywords: Refractive Cataract Extraction; Femtosecond laser; arcuate relaxing incisions; Dry Eye post cataract refraction
MeSH Terms: conditions — Cataract; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study objective is to assess changes in corneal sensation and dry eye signs and symptoms following cataract extraction/femtosecond arcuate relaxing incisions.

Our clinical hypothesis is to determine if a combination of cataract surgery and femtosecond arcuate relaxing incisions lead to a reduction in corneal sensation and the onset or worsening of dry eye signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older, in good general health
* Prior to signing the Institutional Review Board approved Informed Consent Form / Health Insurance Portability and Accountability Act subject read and gained an understanding of the contents
* Subject scheduled for cataract extraction with intraocular lens and requiring two (2) femtosecond arcuate relaxing incisions for correction of corneal astigmatism
* Subject has greater than or equal to 1.0 D and less than or equal to 2.5 Diopters of corneal astigmatism as measured by keratometry or corneal topography
* Two (2) arcuate incisions should be 45° in length and 180° apart.
* All arcuate relaxing incisions will be placed exactly 4.5 mm from the visual axis for a 9 mm optical zone.
* Corneal sensation at Screening by Cochet-Bonnet Aesthesiometry with floor stand >50 mm in all five regions
* Be willing / able to return for all required study visits and comply with instructions given by study staff
* Potential for best corrected visual acuity post cataract surgery of 20/20

Exclusion Criteria:

* Uncontrolled inflammation not related to dry eye
* Corneal abnormality that can affect corneal sensation or tear film stability (except superficial punctate keratitis (SPK)).
* History of ophthalmic herpes simplex or zoster keratitis
* OSDI score > 32
* Active ocular allergy
* History of refractive surgery or any surgery involving conjunctival, arcuate or corneal incision
* Contact lens wear during the study. Soft contact lens wearers should discontinue use at least two weeks prior to Screening visit. Rigid gas permeable (RGP) or hard contact lens wearers should discontinue use at least one month prior to Screening visit.
* Dry eye secondary to Vitamin A deficiency, scarring, pemphigoid, alkali burns, Stevens-Johnson syndrome, trachoma, or irradiation.
* Currently using, or have used within 14 days of study enrollment, any ocular medications other than artificial tears
* Use of topical cyclosporine (Restasis) within three months of Screening visit.
* Have an uncontrolled systemic disease (e.g., hypertension, diabetes) or the presence of any significant illness (e.g., serious gastrointestinal, renal, hepatic, endocrine, pulmonary, cardiac, neurological disease, cancer, AIDS, or cerebral dysfunction) that could, in the judgment of the investigator, jeopardize subject safety or interfere with the interpretation of the results of the study
* Temporary or permanent occlusion of the lacrimal puncta
* Require chronic use of systemic medications which may induce or affect a dry eye condition (e.g., anticholinergics, cyclosporine, antihistamines, antimuscarinics, beta-blocking agents, tricyclic antidepressants, phenothiazines, estrogen-progesterone, and other estrogen derivatives), unless that medication has been used in the same dose for at least 3 months and is expected to remain constant for the course of the study
* Current or anticipated use of nutritional supplements (e.g. flax seed oil, fish oil, omega-3 supplements) which may affect a dry eye condition.
* Are currently enrolled in any other clinical study or have participated in such a study within 30 days of entry into this study
* Is pregnant, breast-feeding, planning a pregnancy, or not using a reliable method of contraception. Subjects who become pregnant during the study will be discontinued from further study participation.
* Have a condition or are in a situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Private Practice
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Sensitivity Testing | Change from Screening to Month 3
  Subject lies supine with the test line of the Cochet-Bonnet Aesthesiometer suspended over the cornea to measure the sensation of touch on the eye. Testing is done in a standard manner by an experienced operator.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Change from Screening to Month 3
  Subject questionnaire
Subject Dry Eye Questionnaire | Change from Screening to Month 3
  Subject questionnaire
Artificial Tear Use | Change from Screening to Month 3
  Subject questionnaire
Corneal and Conjunctival Staining | Change from Screening to Month 3
  Clinical assessment of Dry Eye severity on the cornea via the use of fluorescein dye and on the conjunctiva via the use of lissamine green dye.
Tear Break Up Time (TBUT) with Biomicroscopy | Change from Screening to Month 3
  Clinical assessment of Dry Eye severity via Biomicroscopy with fluorescein dye
Best Corrected Visual Acuity (BCVA) | Change from Screening to Month 3
  Best Corrected Visual Acuity via eye chart examination
Intraocular Pressure (IOP) | Change from Screening to Month 3
  Intraocular pressure via slit lamp examination

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthlamic Consultants of Long Island - Rockville Centre, Rockville Centre, New York, United States